CLINICAL TRIAL: NCT03506958
Title: Patient Satisfaction in Treatment of Non-complex Fractures and Dislocations in Hospitals Versus in General Practitioners in the Netherlands: Prospective Cohort Study Protocol
Brief Title: Patient Satisfaction in Treatment of Non-complex Fractures and Dislocations in Hospitals vs General Practitioners
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Antonius Hospital Sneek (Unknown); Innovatiefonds De Friesland Zorgverzekeraar (DFZ) (Unknown)
Responsible Party: Principal Investigator, dr. T. Verbeek, Post-doc researcher, University Medical Center Groningen
Other Study IDs: 20170277
Record Dates: First submitted 2018-04-07; First posted 2018-04-24 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Fractures, Bone; Dislocations
MeSH Terms: conditions — Fractures, Bone; Joint Dislocations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Practice: Hundred patients with an X-ray confirmed diagnosis of a non-complex fracture or dislocation and planned to be treated in the general practice Zorgplein Lemmer.
  Interventions: Procedure: Standard trauma care
- Hospital: Hundred patients with an X-ray confirmed diagnosis of a non-complex fracture or dislocation and planned to be treated in the Antonius Hospital Sneek.
  Interventions: Procedure: Standard trauma care

INTERVENTIONS:
Procedure: Standard trauma care — In both groups, all procedures and management will be done according to the hospital's standard of care.

SUMMARY:
Treatment of fractures and dislocations are generally organized in the hospital setting. However, equal care for patients with non-complex fractures or dislocations may be provided in general practices. While substitution of trauma care from the secondary to the primary care setting is stimulated by the government and insurers, it is unknown what the patient satisfaction level is and which determinants affect this patient satisfaction. Therefore, the primary objective of this study is to determine the effect of treatment in a general practice on patient satisfaction compared to treatment in a hospital. The secondary objectives include assessments in quality of life, patient-reported outcomes and cost-effectiveness. Besides, results will be discussed using a small focus group consisting of patients (n=15 per group) and healthcare providers.

ELIGIBILITY:
Inclusion Criteria:

* X-ray confirmed diagnosis of a non-complex fracture or dislocation, which can be treated in the primary care setting according to the treatment protocol.
* Ability of the patient or assigned representative to understand the content of the patient information/informed consent form.
* Signed and dated written informed consent. Parents of patients of age 12-17 must provide a signed and dated written informed consent as well.

Exclusion Criteria:

* Patients of age 11 years and younger.
* Patients presenting outside ordinary business hours.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Two hundred patients with an X-ray confirmed diagnosis of a non-complex fracture or dislocation and planned to be treated in either the general practice Zorgplein Lemmer or Antonius Hospital Sneek will be recruited, 100 per center.
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 12 weeks after treatment
  Patient satisfaction measured using the Patient Satisfaction Questionnaire Short Form (PSQ-18)

SECONDARY OUTCOMES:
Patient satisfaction | 1 week and 6 weeks after treatment
  Patient satisfaction measured using the Patient Satisfaction Questionnaire Short Form (PSQ-18)
Complications of treatment | 12 weeks after treatment
  Assessment of treatment complications
Pain score | 12 weeks after treatment
  Assessment of pain score using a visual-analogue scale (VAS)
Physical functioning | 12 weeks after treatment
  Physical functioning according to the 12-item World Health Organisation (WHO) Disability Assessment Schedule II
Limitations in functions of upper extremities (if applicable) | 12 weeks after treatment
  Limitations in functions of upper extremities according to the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire
General health status | 12 weeks after treatment
  General health status according to the General Health Questionnaire (GHQ)
Quality of life | 12 weeks after treatment
  Quality of life using the EuroQol (EQ5D) questionnaire
Time consumption | 1 week, 6 weeks, and 12 weeks after treatment
  Time consumption (waiting time, treatment time, travelling time)
Costs | 12 weeks after treatment
  Costs of treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - General Practice Zorgplein Lemmer, Lemmer, Provincie Friesland
  - Antonius Hospital Sneek, Sneek, Provincie Friesland

REFERENCES:
- [Derived] Verbeek T, Arentsen H, Breet EJ, Kuipers MM, Lubbert PHW, Burger H. Patient satisfaction in treatment of non-complex fractures and dislocations in general practice in the Netherlands: prospective cohort study protocol. BMJ Open. 2019 Feb 19;9(2):e025046. doi: 10.1136/bmjopen-2018-025046. PMID 30782924

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/58/NCT03506958/Prot_SAP_000.pdf